CLINICAL TRIAL: NCT01855386
Title: Non-Alcoholic Fatty Liver Disease in Gestational Diabetes - An Opportunity for Prevention of Type 2 Diabetes Mellitus?
Brief Title: The Role of Non-Alcoholic Fatty Liver Disease in Gestational Diabetes
Status: Terminated | Type: Observational
Why Stopped: Expired with the IRB
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201600437; 375-2012 (Other: University of Florida)
Record Dates: First submitted 2013-03-21; First posted 2013-05-16 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy
MeSH Terms: interventions — Blood Pressure; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with Gestational Diabetes: Subjects with a history of Gestational Diabetes will provide blood samples, blood pressure measured with a blood pressure cuff, pulse, height, weight, and ultrasound of the liver at the 6 week postpartum and 6 month postpartum visits.
  Interventions: Other: Subjects with Gestational Diabetes
- Controls without Gestational Diabetes: Matched control subjects without Gestational Diabetes will provide blood samples, blood pressure measured with a blood pressure cuff, pulse, height, weight, and ultrasound of the liver at the 6 week postpartum and 6 month postpartum visits.
  Interventions: Other: Controls without Gestational Diabetes

INTERVENTIONS:
Other: Subjects with Gestational Diabetes — Subjects with a history of Gestational Diabetes will provide blood samples, blood pressure measured with a blood pressure cuff, pulse, height, weight, and ultrasound of the liver at the 6 week postpartum and 6 month postpartum visits.
  Other Names: Gestational Diabetes; Liver ultrasound; blood pressure; blood samples
  Groups: Subjects with Gestational Diabetes
Other: Controls without Gestational Diabetes — Matched control subjects without gestational diabetes will provide blood samples, blood pressure measured with a blood pressure cuff, pulse, height, weight, and ultrasound of the liver at the 6 week postpartum and 6 month postpartum visits.
  Other Names: Liver ultrasound; blood pressure; blood samples
  Groups: Controls without Gestational Diabetes

SUMMARY:
The thought is that Non-Alcoholic Fatty Liver Disease (NAFLD) plays a key role in the progression to prediabetes/T2DM in those with a history of Gestational Diabetes (GDM). The investigators want to know if having a fatty liver will be connected with more glucose abnormalities (higher fasting/oral glucose tolerance test glucose, more insulin resistance) and that a history of GDM will be common in those with NAFLD.

DETAILED DESCRIPTION:
A liver ultrasound will be completed during the last trimester of pregnancy along with a questionnaire. The questionnaire includes baseline maternal characteristics, age, race, ethnicity, parity, blood pressure, pulse, medications, activity level, sociodemographic and behavioral risk factors, pregravid BMI, previous obstetric history, medical and family history.

The subject will come in person to clinic two times after the subject has had her baby (at 6 weeks postpartum, and at 6 months postpartum).

The subject will give blood samples during the 6 weeks postpartum visit and 6 months postpartum visit, and an Oral Glucose Tolerance Test will be done at these visits. Blood samples will be drawn by putting a small needle or IV catheter (a small plastic tube) into a vein in the subject's arm. Blood samples will be obtained at timed intervals both before and after the subject is given a glucose beverage to drink, to see how well the subject's body deals with sugar in the blood over time. The total amount of blood to be drawn for each Oral Glucose Tolerance Test and research blood work will be approximately 90 ml (about 6 tablespoons). The total volume of blood taken over the course of the study for each subject will be approximately 180 ml (about 12 tablespoons).

The subject will have their blood pressure measured with a blood pressure cuff during each clinic visit. The height, weight and pulse rate will also be measured. This will take about five minutes.

The subject will have an ultrasound of her liver at the 6 week postpartum visit and 6 month postpartum visit. This will take about 30 to 60 minutes each time.

The investigator's study coordinator will call the subject to do a questionnaire over the phone at 3 months after the subject has had the baby. During the phone call, the study coordinator will ask the subject how the baby is being fed. The study coordinator will also update information about development of any new medical problems and medications the subject's doctor might have started, activity levels, and health habits. Subjects will be asked questionnaires to update this information during their 6 week postpartum and 6 month postpartum clinic visits as well.

The subject's understanding and approval of these procedures is required if she is to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* a pregnant female
* age between 18-50 years.

Exclusion Criteria:

* pregravid diabetes mellitus
* inability to understand and speak English
* inability to provide consent
* plans to relocate out of the area within 12 months postpartum

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: * a pregnant female
  * age between 18-50 years.
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with NAFLD and gestational diabetes. | 6 months
  Patients with gestational diabetes will be screened for fatty liver by ultrasound to estimate the prevalence of NAFLD in this population.

SECONDARY OUTCOMES:
Insulin sensitivity expressed as the Matsuda Index, measured during an oral glucose tolerance test (OGTT). | At 6 weeks and 6 months after delivery
  Patients will undergo an OGTT at 6 weeks and 6 months after delivery to measure their insulin sensitivity (which will be expressed as Matsuda Index).

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Sattari, MD, Principal Investigator — University of Florida
Locations (1):
- Shands Medical Plaza, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No